CLINICAL TRIAL: NCT02731300
Title: Transcranial Direct Current Stimulation for Treatment of Childhood Pharmacoresistant Lennox-Gastaut Syndrome, A Pilot Study
Brief Title: Transcranial Direct Current Stimulation, Treatment of Childhood Drug-Resistant Lennox-Gastaut Syndrome, A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Paradee Auvichayapat, Head of Noninvasive Brain Stimulation Research Group of Thailand, Department of Physiology; Faculty of Medicine, Khon Kaen University, Khon Kaen 40002, Thailand., Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: tDCSLennox
Record Dates: First submitted 2016-03-30; First posted 2016-04-07 (Estimated); Results first posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-05

CONDITIONS: Lennox-Gastaut Syndrome
Keywords: Transcranial direct current stimulation; Cathodal stimulation; Childhood Pharmacoresistant epilepsy; Lennox-Gastaut syndrome
MeSH Terms: conditions — Lennox Gastaut Syndrome | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active tDCS (Active Comparator): 2 mA of cathodal tDCS placed over M1 for 20 mins
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): 0 mA of sham tDCS placed over M1 for 20 mins
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — brain stimulation by cathodal electrode at motor cortex

SUMMARY:
Background: Lennox-Gastaut syndrome (LGS) is a severe childhood epileptic syndrome with high pharmacoresistance. The treatment outcomes are still unsatisfied. The investigator previous study of cathodal transcranial direct current stimulation (tDCS) in children with focal epilepsy showed significant reduction in epileptiform discharges. The investigator hypothesized that cathodal tDCS when applied over the primary motor cortex (M1) combined with pharmacologic treatment will be more effective for reducing seizure frequency in participants with LGS than pharmacologic treatment alone.

Material and Method:

Study participants were randomized to receive either:

1. pharmacologic treatment with 5-consecutive days of 2 milliampere (mA) cathodal tDCS over M1 for 20 min or
2. pharmacologic treatment plus sham tDCS. Measures of seizure frequency and epileptic discharges were performed before treatment and again immediately post-treatment and 1-, 2-, 3-, and 4-week follow-up.

DETAILED DESCRIPTION:
Participant recruitment and informed consent Study participants were recruited via advertisement at the pediatric outpatient department, Srinagarind Hospital, Faculty of Medicine, Khon Kaen University, Thailand. The study procedures were described to any eligible participants who expressed an interest in participating in the study by a pediatric neurologist.

Criteria for LGS were defined according to the triad of:

1. polymorphic intractable seizures that are mainly tonic, atonic, and atypical absence seizures,
2. cognitive and behavioral abnormalities,
3. EEG with paroxysms of fast activity and slow (less than 2.5 Hz) generalized spike-wave discharges (GSWD).

The diagnosis was confirmed by a pediatric neurologist using the thoroughly history taking, physical examination, EEG, and brain MRI.

Study inclusion criteria included:

1. diagnosis of LGS;
2. failure of more than two first-line antiepilepsy drug (AEDs) to control seizures;
3. average seizure frequency of more than one per month for 18 months and no more than three consecutive seizure-free months during that interval;
4. age between 6 and 15 years.

The exclusion criteria were

1. drug addiction, pregnancy, skull defect, and other serious neurological diseases; and
2. change in dosage of antiepileptic drugs or use of herbal remedies and other alternative therapies.

All participants' guardians gave their written informed consent. The study conformed to the declaration of Helsinki and was approved by the Ethics Committee of Khon Kaen University (Identifier number: Human Ethic (HE) 521232.

Experimental design

The current study was a randomized double-blind controlled trial performed over a total of 6 weeks consisting of:

1. a 1-week period of observation to assess the baseline seizure frequency,
2. a 5 consecutive days of 2 mA cathodal tDCS for 30 minutes, and
3. 4 weeks of follow-up.

Just before the treatment phase, study participants were randomized in a 2:1 ratio in blocks of four randomization to receive either (a) pharmacologic treatment plus active tDCS stimulation or (b) pharmacologic treatment plus sham tDCS stimulation for 5 days. Participants were asked to continue their routine anti-epileptic medication regimen throughout the duration of the 6-week trial.

Pharmacologic treatment

Since there is a considerable degree of heterogeneity with LGS, individualized approaches are necessary. The investigator firstly uses the antiepileptic drugs that currently approved by the Food and Drug Administration and available in our institute: lamotrigine, topiramate, clobazam, and clonazepam depended on seizure types. The investigator gave lamotrigine 1-20 mg/kg/day with slowly titration for tonic, tonic-clonic, atypical absences, and atonic seizures. Clobazam 0.25-3.5 mg/kg/day was added in the cases that refractory to lamotrigine and in the participants with myoclonic seizures. The investigator used clonazepam 0.04-0.2 mg/kg/day instead of clobazam in some cases when clobazam was not available. We used topiramate 1-10 mg/kg/day in the participants who refractory to lamotrigine and clobazam. In some cases, that refractory to the aforementioned antiepileptic drugs, the investigator gave zonisamide 1-20 mg/kg/day, levetiracetam 10-80 mg/kg/day, and nitrazepam 0.1-0.8 mg/kg/day [8].

Randomization and Blinding Prior to the treatment phase, study participants were randomized in a 2 : 1 ratio in blocks of four randomizations (by OT) to receive either (1) active tDCS stimulation or (2) sham tDCS stimulation. Participants were asked to continue their routine medication regimen throughout the trial. The staff who generated the random allocation sequence, enrolled participants, and assigned participants to interventions were not involved in any assessments. After assignment to the intervention groups, the pediatric neurologist who carried out the seizure assessments (NA) was blind to treatment condition. Because the study participants were also blind to treatment condition, this is a double-blind study.

Active and Sham Transcranial Direct Current Stimulation.

tDCS was applied via water-soaked pair of surface sponge electrodes (35 cm2) and delivered through battery-driven power supply. The constant current stimulator had a maximum output of 10 mA (Soterixmedical, Model 1224-B, New York, USA). The stimulation site over the left M1, located based on the international electroencephalography (EEG) 10/20 electrode placement system. The reference electrode was placed over the right shoulder area. The tDCS device was designed to allow sham stimulation by placing the control switch in front of the instrument which was easily covered by an opaque adhesive during stimulation. Therefore the participants or their gradients could not know whether active or sham stimulation. The power lit up indicator was also on the front of the machine during the time of intervention both in active and sham stimulations. However, in sham stimulation, the current was discontinued after 30 seconds while the power indicator remained on [18].

Measures Number of seizures Since Lennox-Gastaut Syndrome compose of many seizure types. All seizures were classified according to the International League Against Epilepsy Revised Classification of Seizures [29]. The participants were monitored by video-EEG in order to classify the types and frequencies of seizures, and all of the caregivers were taught how to count and classify seizures on the basis of observations and video recordings. The caregivers were also taught the rules for diary recording prior to the baseline period. All of the caregivers were blinded to both treatment and sham group. In case of the participant who had more than 1 caregiver. The investigator suggested them to refer the daily diary to the person who cared the participant in time.

Number of seizure was the primary outcome variable, and was assessed by using a daily diary. For the baseline (pre-treatment) assessment, the caregivers were asked to record the number of seizures every day for 7 days during the baseline period on a daily diary. These 7 days numbers of seizures were averaged into a single rate per day of baseline average seizure frequency. During the 5 consecutive day of treatment, the caregivers were asked to record the daily children seizure frequency. Finally, daily 24-hour recording were administered for four weeks following treatment. 1-, 2-, 3-, and 4-week composite number of seizures were computed as an average of the daily number of seizures for each epoch (i.e., the 1-week follow-up average number of seizures = average of 7 daily number of seizures the first week after treatment).

Epileptic discharges

Epileptic discharges, the secondary outcome variable of this study, were recorded by a trained staff. EEG was acquired from all participants using a 32-channel, international 10-20 system of electrode placement (Neuvo, Compumedics, Australia with PerFusion EEG software). EEG was collected for 30 minutes in the awake state only. EEG was recorded as a single session at baseline, immediately, 1-, 2-, 3- and 4- weeks follow-ups. EEG data were analyzed by visual inspection. The numbers of epileptic discharges in the 30-minute recording were assessed by a practicing pediatric neurologist and clinical neurophysiologist (N.A.), who was blinded to the treatment condition. The EEGs that included as abnormal EEGs in LGS are slow spike-wave complexes at <3 Hz that occur during wakefulness. The complexes consist of a spike (duration < 70 msec) or a sharp wave (70-200 msec), followed first by a positive deep trough, and then a negative wave (350-400 msec). Paroxysmal fast rhythms (10-20 Hz) occur mainly during non-rapid eye movement sleep [30]. One slow spike-wave complex or one episode of paroxysmal fast rhythms were counted as one epileptic discharge.

Vital signs and oxygen saturation monitoring

All participants were closely observed by physicians during and post-treatment. Oxygen saturation and vital signs were monitored for 30 minutes before, during, and 30 minutes after the treatment. Pulse rate was measured by automatic sphygmomanometer (Ua-767 Plus, UK) in the supine position. Blood pressure (mm Hg) was measured by automatic sphygmomanometer (Ua-767 Plus, UK) in the supine position with a pediatric-size cuff wrapped around the right upper arm. Body temperature was measured by an axillary electronic thermometer. Respiratory rate was measured by counting chest rising for 60 seconds. Pulse oximeter was placed on the left index finger to monitor oxygen saturation throughout the procedure.

Adverse events

Adverse events as well as other signs and symptoms were reported by participants' guardians every day after treatment. Theses self-recordings terminated at 4 weeks after stimulation.

Statistical analysis

The investigator first computed means and standard deviations (SD) of the demographic and outcome variables for descriptive purposes. Next, the investigator compared the two treatment conditions (active tDCS versus sham tDCS) on all baseline outcome measures to ensure baseline equivalence using t-tests. Results are presented as means and SD. Both the primary (seizure frequency) and exploratory (epileptic discharges) hypotheses were tested using repeated measures analysis of variance (ANOVA) followed by Least Significant Difference to help understand any significant effects found. To describe the clinically meaningfulness of any changes, the investigator computed the percent reduction of number of seizures and epileptic discharges in each condition from pre- to post-treatment and from pre-treatment to 4-week follow-up. For all analyses, p values of < 0.05 were considered statistically significant. Analyses were completed using STATA software, version 10.0 (StataCorp, College Station, TX).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of LGS
* Failure of more than two first-line AEDs to control seizures
* Average seizure frequency of more than one per month for 18 months and no more than three consecutive seizure-free months during that interval
* Age between 6 and 15 years

Exclusion Criteria:

* Drug addiction
* Pregnancy
* Skull defect
* Other serious neurological diseases and change in dosage of antiepileptic drugs or use of herbal remedies and other alternative therapies.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2010-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Auvichayapat N, Sinsupan K, Tunkamnerdthai O, Auvichayapat P. Transcranial Direct Current Stimulation for Treatment of Childhood Pharmacoresistant Lennox-Gastaut Syndrome: A Pilot Study. Front Neurol. 2016 May 4;7:66. doi: 10.3389/fneur.2016.00066. eCollection 2016. PMID 27199889

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited via advertisement at the pediatric outpatient department, Srinagarind hospital, Faculty of Medicine, Khon Kaen University, Thailand. A total of 22 patients with Lennox-Gastaut Syndrome (LGS) were enrolled between August 2010 and December 2013
Pre-assignment Details: All patients were assigned to record sizure frequency prior to start the protocol
Groups:
- Active tDCS: 2 milliampere (mA) of cathodal tDCS placed over M1 for 20 mins
  tDCS: brain stimulation by cathodal electrode at motor cortex
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 15 | 7
Completed | 15 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 15 | 7 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.67 (1.54) | 6.29 (1.98) | 6.55 (1.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 9 | 5 | 14
Etiologies of epilepsy [Number; unit: participants]
  Idiopathic | 6 | 2 | 8
  Infantile spasm | 1 | 1 | 2
  Neonatal hypoglycemia | 4 | 3 | 7
  Preterm with severe birth asphyxia | 2 | 0 | 2
  Preterm with history of intercerebral hemorrhage | 2 | 1 | 3
Baseline seizure frequency per day [Mean (Standard Deviation); unit: seizures per day] | 80.67 (54.43) | 93.43 (59.94) | 84.73 (55.13)
Baseline epileptic discharges per 30 minutes [Mean (Standard Deviation); unit: epileptic discharges/30 mins] | 640.13 (263.30) | 800.86 (374.62) | 691.27 (303.62)
Age at onset of seizures [Mean (Standard Deviation); unit: years] | 2.32 (2.39) | 1.58 (1.70) | 2.08 (2.18)
Number of antiepileptic drugs used [Number; unit: participants]
  3 drugs | 9 | 3 | 12
  4 drugs | 4 | 2 | 6
  5 drugs | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Seizure After Treatment by tDCS
Time Frame: Baseline, 4 Weeks
Measure: Mean (Standard Deviation); unit: seizures
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 15 | 7
seizures
  Baseline | 80.67 (54.43) | 93.43 (59.95)
  Week4 | 35.53 (15.29) | 93.14 (61.15)
Statistical Analysis 1: Comparison: Active tDCS vs Sham tDCS; the final Week 4 values compared between active tDCS and sham tDCS groups; Test type: Superiority or Other; p < 0.05, ANOVA — the final Week 4 values compared between active tDCS and sham tDCS groups

2. Secondary Outcome: Number of Epileptic Discharge After Treatment by tDCS
Time Frame: Baseline, 4 Weeks
Measure: Mean (Standard Deviation); unit: epileptic discharges/30 mins
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 15 | 7
epileptic discharges/30 mins
  Baseline | 640.13 (263.30) | 800.86 (374.62)
  Week4 | 585.33 (253.25) | 831.43 (392.22)
Statistical Analysis 1: Comparison: Active tDCS vs Sham tDCS; the final Week 4 values compared between active tDCS and sham tDCS groups; Test type: Superiority or Other; p < 0.05, ANOVA — the final Week 4 values compared between active tDCS and sham tDCS groups

ADVERSE EVENTS:
Arm/Group | Active tDCS | Sham tDCS
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/7
Other Adverse Events (participants affected / at risk) | 1/15 | 0/7
OTHER ADVERSE EVENTS (reported when occurring in more than 4.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active tDCS (N=15) | Sham tDCS (N=7)
superficial skin burn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — superficial skin burn under the reference electrode in active tDCS group, which resolved within 2 days.

LIMITATIONS AND CAVEATS:
1. The investigators could not ensure that the stimulation electrode was directly over the primary motor cortex.
2. The sample size was small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No